CLINICAL TRIAL: NCT04478500
Title: The Role of Neuroinflammation in Hypertension.Minocycline for Resistant Hypertension: a Randomized Double Blind Placebo-Controlled Trial
Brief Title: Neuroinflammation in Hypertension Study
Acronym: MINIHT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Perth Hospital (Other)
Responsible Party: Principal Investigator, Dr Markus Schlaich, Professor, Royal Perth Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DHC20180023
Record Dates: First submitted 2020-07-10; First posted 2020-07-20 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Resistant Hypertension
MeSH Terms: interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minocycline Group (Active Comparator): Subjects will be randomized to receive Minocycline 100mg twice daily
  Interventions: Drug: Minocycline
- Placebo Group (Placebo Comparator): Subjects will be randomized to receive placebo.
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Participants will be randomly assigned to receive either Minocycline 100mg twice daily or Placebo.
  Comprehensive testing will be performed at baseline, and at the end of the 12 week intervention phase.
  Other Names: Akamin

SUMMARY:
To demonstrate that in patients with resistant hypertension oral treatment with minocycline via inhibition of central immune cell activation and inflammation results in reduced central sympathetic outflow and concomitant lowering of BP.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, parallel group design study aiming to compare the effects of minocycline 100mg twice daily vs matched placebo for 12 weeks on ambulatory BP and the parameters of sympathetic and immune activation

ELIGIBILITY:
Inclusion Criteria:

* Aged: 45 -65 years
* Signed informed consent
* Clinical diagnosis of Resistant Hypertension
* Daytime systolic ambulatory BP >135mmHg.

Exclusion Criteria:• eGFR of <45 mL/min/1.73m2

* History of myocardial infarction (MI) or any cardiovascular event within 3 months of screening period, clinically significant AV conduction disturbances and/or arrhythmias,
* current of past history of heart failure (LVEF ≤40%)
* psychotropic agents, antidepressants and NSAIDS
* alcohol consumption of >3 standard drinks.
* known hypersensitivity or contraindication to minocycline or other tetracyclines.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
The difference in the daytime systolic blood pressure between groups after respective treatment. | 12 weeks
  Office and ambulatory blood pressures
Assessment of change in central and peripheral inflammation | 12 weeks
  FDG PET

SECONDARY OUTCOMES:
Change in muscle sympathetic nerve activity | 12 weeks
  Muscle sympathetic nerve activity assessed by microneurography
Change in central Blood Pressure | 12 weeks
  central Blood Pressure assessed by Sphygmocor XCEL

CONTACTS AND LOCATIONS:
Overall Officials: Markus Schlaich, MD, Principal Investigator — University of Western Australia and Royal Perth Hospital
Locations (1):
- Royal Perth Hospital, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carnagarin R, Matthews V, Zaldivia MTK, Peter K, Schlaich MP. The bidirectional interaction between the sympathetic nervous system and immune mechanisms in the pathogenesis of hypertension. Br J Pharmacol. 2019 Jun;176(12):1839-1852. doi: 10.1111/bph.14481. Epub 2018 Sep 25. PMID 30129037
- [Background] Santisteban MM, Ahmari N, Carvajal JM, Zingler MB, Qi Y, Kim S, Joseph J, Garcia-Pereira F, Johnson RD, Shenoy V, Raizada MK, Zubcevic J. Involvement of bone marrow cells and neuroinflammation in hypertension. Circ Res. 2015 Jul 3;117(2):178-91. doi: 10.1161/CIRCRESAHA.117.305853. Epub 2015 May 11. PMID 25963715